CLINICAL TRIAL: NCT05562089
Title: Drug-Coated Balloon for the Treatment of De Novo and Restenotic Coronary Artery Lesion: a Prospective Observational Study
Brief Title: Prevail Drug Balloon Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021.637
Record Dates: First submitted 2022-09-20; First posted 2022-09-30 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Infarction; Drug-Coated Balloon
Keywords: Drug-Coated Balloon; De Novo; Restenotic Coronary Artery Lesion; major adverse cardiac event; target-lesion revascularization; Myocardial infraction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevail (Experimental)
  Interventions: Device: A Paclitaxel Drug-Coated Balloon

INTERVENTIONS:
Device: A Paclitaxel Drug-Coated Balloon — Size: 2.0mm-4.0mm x 15-30mm Coated drug: Prevail TM

SUMMARY:
This is an investigator-initiated, prospective, single-centre, non-randomized, all-comers registry that evaluates the safety and efficacy of any Paclitaxel Drug-Coated Balloon (DCB) for the treatment of coronary de novo lesion, in-stent restenosis, and small vessel disease in patients with coronary artery disease in Hong Kong. The recruitment time frame of this study is 1 year from 1st January 2022 to 30th December 2022.

DETAILED DESCRIPTION:
Procedural strategy, adjuvant medical therapy and antiplatelet regime were left to the discretion of individual operators and their routine clinical practice. In brief, lesion preparation with predilatation using an uncoated balloon with or without the use of adjunctive therapy such as atherectomy or intracoronary lithotripsy to achieve residual diameter stenosis of less than 30% will be required before the usage of the study device. If the lesion meets the inclusion criteria without any of the exclusion criteria, the DCB of appropriate diameter and length can be applied with a minimum inflation time of 30-60 seconds. More than 1 lesion can be treated using the study device in the same vessel. Bail-out stenting is allowed as per operators' discretion.

Baseline demographic, clinical and angiographic characteristics of each patient will be recorded. Both 6 and 12 months clinical outcomes and procedural outcomes will be assessed. Patient will be reviewed by the treating physicians before discharge and at clinic as per local practice. The primary clinical endpoint is the 12 months major adverse cardiac event (MACE), defined as a composite of death, Myocardial infraction (Q-wave and non-Q wave), emergent coronary artery bypass graft surgery, or repeat clinically driven target-lesion revascularization (TLR) by percutaneous or surgical methods. The primary procedural outcomes are device success which defined as achieving less than 50% residual stenosis after the usage of only the study device, the lesion success defined as achieving less than 50% residual stenosis of target lesion using any percutaneous method, and procedural success, defined as lesion success and no in-hospital MACE during the index admission.

Categorical variables will be reported as percentages and counts, and continuous variables will be reported as means ± standard deviations. Data analysis will be performed using STATA version 15 software (College Station, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

1. Subject age >18.
2. Subject (or legal guardian) understands the trial requirements and treatment procedures and provides written informed consent prior to any trial-specific tests or treatment.
3. Indication for a percutaneous intervention in native epicardial arteries or bypass graft including patients with stable coronary artery disease and acute coronary syndromes (non- ST-elevated myocardial infarction and ST-elevation myocardial infarction).
4. Target lesion must have a stenosis of >50% and <100% angiographically.
5. Target lesion much have an angiographic reference vessel diameter of 2.0-4.0 mm.
6. Successful predilatation of the target lesions as defined by angiographic visual estimate of <30% residual stenosis without major (defined as >NHLBI grade B) flow-limiting dissection.
7. Target lesion must have a Thrombolysis in Myocardial Infarction flow >2 before applying DCB.

Exclusion Criteria:

1. Known history of an allergic reaction or significant sensitivity to paclitaxel or other analogue or derivative.
2. Known history of an allergic reaction or significant sensitivity to urea or its analogue or derivative.
3. Pregnant or breastfeeding woman.
4. Currently participating in an investigational drug or another device study that has not completed the primary end point or that clinically interferes with the current study endpoints.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE) | 12 month
  Major adverse cardiac events (MACE) were defined as the composite of total death; myocardial infraction; stroke, hospitalization because of heart failure; and revascularization, including percutaneous coronary intervention, and coronary artery bypass graft
Device success | 12month
  device success which defined as achieving less than 50% residual stenosis after the usage of only the study device
Lesion success | 12 month
  the lesion success defined as achieving less than 50% residual stenosis of target lesion using any percutaneous method
Procedural success | 12 month
  the procedural success defined as lesion success and no in-hospital MACE during the index admission

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Result] Byrne RA, Joner M, Kastrati A. Stent thrombosis and restenosis: what have we learned and where are we going? The Andreas Gruntzig Lecture ESC 2014. Eur Heart J. 2015 Dec 14;36(47):3320-31. doi: 10.1093/eurheartj/ehv511. Epub 2015 Sep 28. PMID 26417060
- [Result] Stone GW, Kimura T, Gao R, Kereiakes DJ, Ellis SG, Onuma Y, Chevalier B, Simonton C, Dressler O, Crowley A, Ali ZA, Serruys PW. Time-Varying Outcomes With the Absorb Bioresorbable Vascular Scaffold During 5-Year Follow-up: A Systematic Meta-analysis and Individual Patient Data Pooled Study. JAMA Cardiol. 2019 Dec 1;4(12):1261-1269. doi: 10.1001/jamacardio.2019.4101. PMID 31561250
- [Result] Chien S. Mechanotransduction and endothelial cell homeostasis: the wisdom of the cell. Am J Physiol Heart Circ Physiol. 2007 Mar;292(3):H1209-24. doi: 10.1152/ajpheart.01047.2006. Epub 2006 Nov 10. PMID 17098825
- [Result] Gyongyosi M, Yang P, Khorsand A, Glogar D. Longitudinal straightening effect of stents is an additional predictor for major adverse cardiac events. Austrian Wiktor Stent Study Group and European Paragon Stent Investigators. J Am Coll Cardiol. 2000 May;35(6):1580-9. doi: 10.1016/s0735-1097(00)00570-2. PMID 10807464
- [Result] Latib A, Colombo A, Castriota F, Micari A, Cremonesi A, De Felice F, Marchese A, Tespili M, Presbitero P, Sgueglia GA, Buffoli F, Tamburino C, Varbella F, Menozzi A. A randomized multicenter study comparing a paclitaxel drug-eluting balloon with a paclitaxel-eluting stent in small coronary vessels: the BELLO (Balloon Elution and Late Loss Optimization) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2473-80. doi: 10.1016/j.jacc.2012.09.020. Epub 2012 Nov 14. PMID 23158530
- [Result] Basavarajaiah S, Latib A, Shannon J, Naganuma T, Sticchi A, Bertoldi L, Costopoulos C, Figini F, Carlino M, Chieffo A, Montorfano M, Colombo A. Drug-eluting balloon in the treatment of in-stent restenosis and diffuse coronary artery disease: real-world experience from our registry. J Interv Cardiol. 2014 Aug;27(4):348-55. doi: 10.1111/joic.12129. Epub 2014 May 11. PMID 24815951
- [Result] Widder JD, Cortese B, Levesque S, Berliner D, Eccleshall S, Graf K, Doutrelant L, Ahmed J, Bressollette E, Zavalloni D, Piraino D, Roguin A, Scheller B, Stella PR, Bauersachs J. Coronary artery treatment with a urea-based paclitaxel-coated balloon: the European-wide FALCON all-comers DCB Registry (FALCON Registry). EuroIntervention. 2019 Jul 20;15(4):e382-e388. doi: 10.4244/EIJ-D-18-00261. PMID 29992902
- [Result] Latib A, Agostoni P, Dens J, Patterson M, Lancellotti P, Tam FCC, Schotborgh C, Kedhi E, Stella P, Shen C, Wetzels G, Testa L; PREVAIL Study Investigators. Paclitaxel Drug-Coated Balloon for the Treatment of De Novo Small-Vessel and Restenotic Coronary Artery Lesions: 12-Month Results of the Prospective, Multicenter, Single-Arm PREVAIL Study. J Invasive Cardiol. 2021 Nov;33(11):E863-E869. doi: 10.25270/jic/21.00119. Epub 2021 Aug 19. PMID 34433695